CLINICAL TRIAL: NCT06784414
Title: Analysis of Risk Factors for Recurrence of Periprosthetic Infection in Megaprostheses Implanted for Sarcoma of Bone
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MEGAINF
Record Dates: First submitted 2024-11-28; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: PJI
Keywords: megaprosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to collect a large and homogeneous case report of periprosthetic infections in megaprostheses in patients with a history of bone sarcoma.

DETAILED DESCRIPTION:
The incidence of periprosthetic infections (PJI) is high in megaprostheses (MP), 3-30% after primary surgery, up to 60% after prosthetic revision. Patients with megaprosthesis implanted in a primary sarcoma of bone have an increased risk of infection, compared with joint prostheses implanted on arthrosis, due to several factors, including treatment with chemotherapy, extensive periarticular soft tissue sacrifice, and duration of surgery. PJI of an MP can result in important consequences: prolonged hospitalizations, expensive treatments, multiple surgeries, risk of amputation and reduced quality of life.

Diagnosis and treatment of MP infections are challenging. Surgery is the focus of treatment, and identification of the microorganism responsible for infection is necessary for diagnostic confirmation and to set up targeted antibiotic treatment.

Treatment, similar to standard joint replacement, includes surgical cleaning without implant replacement and complete revision of the prosthesis in one or two stages. Data currently available in the Literature about patients with infection of a megaprosthesis implanted after excision of a bone sarcoma is scarce; in particular, most case series are small and heterogeneous.

The aim of this study is to obtain more information about this condition by collecting a large and homogeneous data of PJI in MP, in order to identify predictive factors in the treatment of PJI.

The treatments to which the patients underwent and thus analyzed for the study are those expected by normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PJI caused by a megaprosthesis, implanted for a primary sarcoma of bone;
* Age >= 18 years at the time of diagnosis;
* Megaprosthesis site: proximal humerus, proximal femur, total femur, distal femur, tibia proximal;
* Prosthetic revision in two stages;
* Obtaining informed consent for the study

Exclusion Criteria:

* Early infection (within 6 weeks after implantation of the prosthesis);
* Recurrence of infection;
* Follow-up < 12 months after prosthetic re-implantation;
* Reconstruction other than a megaprosthesis (e.g., bone graft, composite prosthesis)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants meeting the inclusion criteria, processed from 2010 to 2020, were included.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of predictive factors for infection recurrence in patients with PJI: analysis of demographic, prognostic and treatment data. | Data covering the period 2010-2020.
  Demographic information on disease definition, prognosis, treatments provided and outcomes will be summarised using descriptive methods. treatments provided and outcomes, will be summarised using descriptive methods. In in particular, categorical variables will be summarised by means of relative frequency estimation and 95% confidence intervals; continuous variables will be summarised by means of mean and standard deviation, median and range. standard deviation, median and interquartile range.
  Correlations between variables will be investigated: by means of contingency tables and calculation of the chi-square calculation (applying correction for continuity and/or exact test when necessary) for categorical categorical variables; comparison of means (t-test for paired and unpaired data or non-parametric analogues non-parametric when indicated) for variables distributed on an interval scale.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sambri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - A.O.U Città della Salute e della Scienza di Torino, Torino